CLINICAL TRIAL: NCT00532974
Title: A Phase 1 Safety and Immunogenicity Study of the Pharmexa-Epimmune HIV-1 CTL Epitope-Based DNA Vaccine (EP HIV-1090) Administered Using a Biojector 2000 Needle Free Immunization Device in HIV-1 Infected Individuals Receiving Potent Combination Antiretroviral Therapy (ART)
Brief Title: A Phase 1 Safety and Immunogenicity Study of the Epitope Based DNA Vaccine (EP HIV-1090) in HIV-1 Infected Individuals Receiving Antiretroviral Therapy (ART)
Acronym: EP1090
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Epimmune (Industry)
Collaborators: Pharmexa A/S (Industry); Pharmexa-Epimmune (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EP-HIV-1090
Record Dates: First submitted 2007-09-19; First posted 2007-09-21 (Estimated); Last update posted 2007-12-24 (Estimated); Status verified 2007-12

CONDITIONS: HIV Infections
Keywords: HIV; Human Immunodeficiency Virus; Vaccines; HIV Vaccines; Peptide; Peptide Vaccines; HIV 1
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: EP1090 — Low dose
Biological: EP1090 — High dose

SUMMARY:
The use of a Bioject 2000 needle free injection device (NFID) and a compressed immunization schedule will be safely tolerated and will augment the immunogenicity of the HIV-1 CTL epitope DNA vaccine (EP1090) in HIV-1 infected individuals receiving potent combination antiretroviral therapy (ART) and who have undetectable levels of viral replication in plasma.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 Infection
* CD4 Tcell count >350
* HIV-1 RNA levels to <400 copies
* Negative HbsAg and anti-HCV antibody

Exclusion Criteria:

* Recent receipt of experimental HIV-1 vaccines
* Recent use of immunomodulatory agents
* Hypersensitivity or serious reactions to study vaccine components
* Active opportunistic infections

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2006-10; Study Completion 2008-04 (Estimated)

PRIMARY OUTCOMES:
Safety and Immunogenicity: defined as the effect of the vaccine on peripheral blood CD8 CTL responses, CD4 T cell counts, plasma HIV-1 RNA levels and clinical signs and symptoms. | six months

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - AIDS Research Alliance, West Hollywood, California
  - University of Colorado Health Sciences Center, Denver, Colorado